CLINICAL TRIAL: NCT00950339
Title: Platelet Inhibitory Effect of Clopidogrel in Patients Treated With Omeprazole, Pantoprazole, or Famotidine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Tel Aviv Medical Center (Other)
Responsible Party: Principal Investigator, michal roll, Interventional cardiologist, Tel-Aviv Sourasky Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-09-SB-0196-09-TLV-CTIL
Record Dates: First submitted 2009-04-19; First posted 2009-07-31 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Heart Disease; GI Bleeding
Keywords: GI bleeding; clopidogrel; aspirin; prevention; angiography
MeSH Terms: conditions — Coronary Disease; Gastrointestinal Hemorrhage | interventions — Omeprazole; Famotidine; Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 4 weeks of omeprazole, 20mg twice daily (Experimental): Each patient will undergo 3 phases of drug therapy:
  A- 4 weeks of PPI treatment (omeprazole, 20mg twice daily)) B- 4 weeks of H2 blocker treatment (famotidine 40mg twice daily) C- 4 weeks of PPI treatment (pantoprazole 40mg once daily).
  At the end of each phase- each patient will undergo the following evaluation:
  Platelet reactivity
  Interventions: Drug: omeprazole, 20mg twice daily; Drug: famotidine 40mg twice daily; Drug: pantoprazole 40mg once daily
- 4 weeks of famotidine 40mg twice daily (Experimental): Each patient will undergo 3 phases of drug therapy:
  A- 4 weeks of PPI treatment (omeprazole, 20mg twice daily)) B- 4 weeks of H2 blocker treatment (famotidine 40mg twice daily) C- 4 weeks of PPI treatment (pantoprazole 40mg once daily).
  At the end of each phase- each patient will undergo the following evaluation:
  Platelet reactivity
  Interventions: Drug: omeprazole, 20mg twice daily; Drug: famotidine 40mg twice daily; Drug: pantoprazole 40mg once daily
- 4 weeks of pantoprazole 40mg once daily (Experimental): Each patient will undergo 3 phases of drug therapy:
  A- 4 weeks of PPI treatment (omeprazole, 20mg twice daily)) B- 4 weeks of H2 blocker treatment (famotidine 40mg twice daily) C- 4 weeks of PPI treatment (pantoprazole 40mg once daily).
  At the end of each phase- each patient will undergo the following evaluation:
  Platelet reactivity
  Interventions: Drug: omeprazole, 20mg twice daily; Drug: famotidine 40mg twice daily; Drug: pantoprazole 40mg once daily

INTERVENTIONS:
Drug: omeprazole, 20mg twice daily — Each patient will undergo 3 phases of drug therapy:
  A- 4 weeks of PPI treatment (omeprazole, 20mg twice daily)) B- 4 weeks of H2 blocker treatment (famotidine 40mg twice daily) C- 4 weeks of PPI treatment (pantoprazole 40mg once daily).
  At the end of each phase- each patient will undergo the following evaluation:
  Platelet reactivity
  Other Names: PPI Platelet Inhibitory
Drug: famotidine 40mg twice daily — Each patient will undergo 3 phases of drug therapy:
  A- 4 weeks of PPI treatment (omeprazole, 20mg twice daily)) B- 4 weeks of H2 blocker treatment (famotidine 40mg twice daily) C- 4 weeks of PPI treatment (pantoprazole 40mg once daily).
  At the end of each phase- each patient will undergo the following evaluation:
  Platelet reactivity
  Other Names: PPI Platelet Inhibitory
Drug: pantoprazole 40mg once daily — Each patient will undergo 3 phases of drug therapy:
  A- 4 weeks of PPI treatment (omeprazole, 20mg twice daily)) B- 4 weeks of H2 blocker treatment (famotidine 40mg twice daily) C- 4 weeks of PPI treatment (pantoprazole 40mg once daily).
  At the end of each phase- each patient will undergo the following evaluation:
  Platelet reactivity
  Other Names: PPI Platelet Inhibitory

SUMMARY:
Current guidelines recommend the addition of proton pump inhibitors (PPI) to patients taking double anti-platelet therapy (Aspirin and Clopidogrel) to prevent upper GI bleeding1. Many post percutaneous coronary intervention (PCI) patients are treated with dual anti-platelet medications as well as PPI to prevent upper GI bleeding.

Recently, it was shown that PPI interact with the P450 system in the liver and reduce the platelet inhibitory effect of Clopidogrel2,3. Clopidogrel is activated by CYP2C19, which also metabolizes PPI4. Furthermore, a recent article showed increased mortality in patients taking PPI and clopidogrel compared with patients taking clopidogrel without PPI protection5. The degree of reduction in the platelet inhibitory properties of clopidogrel might vary among the different PPI4.

The use of PPI for GI protection in patients treated with dual anti-platelet therapy is not based on randomized trials, but rather on expert opinion. Since H2 blockers are also effective in preventing acid secretion and are not known to interact with the P450 system that affects clopidogrel, the investigators hypothesized that these group of drugs will not interfere with the positive antiplatelet effects of clopidogrel and therefore will offer a good alternative treatment option.

DETAILED DESCRIPTION:
In this study we will compare 3 different anti-acids regimens and their effect on platelet function

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old.
2. Subject is willing to comply with pre-specified follow-up evaluation and can be contacted by telephone.
3. Use of Clopidogrel (>=75mg) and Aspirin(>=75mg) for at least 1 month.

Exclusion Criteria:

1. Known allergy to PPI of H2 blockers
2. Known thrombocytopenia or thrombocytopathia
3. Subject is currently enrolled in another investigational study of a new drug, biologic or device at the time of study screening. NOTE: Subjects who are participating in the long term follow-up phase of a previously investigational and now FDA-approved product are not excluded by this criterion.
4. Subject with symptomatic heart failure of LVEF ≤ 25%
5. Acute myocardial infarction within the past 30 days.
6. No acute inflammatory event during the past month (e.g. infection, autoimmune or acute coronary event)
7. Concurrent medical condition with a life expectancy of less than 12 months.
8. Known severe renal failure (serum creatinine level >2.5 mg/dl).
9. History of bleeding diathesis or coagulopathy or inability or unwillingness to receive blood transfusions.
10. Evidence of active gastrointestinal bleeding or a history of such bleeding that is not known to have been treated and proven to have resolved.
11. History of hepatitis (viral, ischemic or chemically-induced); clinical jaundice, history of cirrhosis.
12. Patient treated with anticoagulant medication (Coumadin, LMWH)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-08; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Platelet function as assessed by a CPA system | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Banai, MD, Study Chair — Tel Aviv Medical Center, Israel
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arbel Y, Birati EY, Finkelstein A, Halkin A, Kletzel H, Abramowitz Y, Berliner S, Deutsch V, Herz I, Keren G, Banai S. Platelet inhibitory effect of clopidogrel in patients treated with omeprazole, pantoprazole, and famotidine: a prospective, randomized, crossover study. Clin Cardiol. 2013 Jun;36(6):342-6. doi: 10.1002/clc.22117. Epub 2013 Apr 29. PMID 23630016